CLINICAL TRIAL: NCT00599430
Title: Probiotics and Effects on Illness-Related Symptoms for Pre-School Age Children
Brief Title: Evaluation of Probiotics on Symptoms of Upper Respiratory Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danisco (Industry)
Responsible Party: Gregory Leyer / Probiotic Technical Director, Danisco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Danisco - Mao; 06-02-D-011
Record Dates: First submitted 2008-01-03; First posted 2008-01-23 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2008-01

CONDITIONS: Healthy
Keywords: Probiotic; Lactobacillus; NCFM; Bifidobacterium; Healthy children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- Active 1 (Active Comparator): One probiotic strain
  Interventions: Dietary Supplement: Lactobacillus acidophilus NCFM
- Active 2 (Active Comparator): Blend of two strains
  Interventions: Dietary Supplement: Combination of Lactobacillus acidophilus and Bifidobacterium lactis

INTERVENTIONS:
Dietary Supplement: Placebo — Inert excipient
  Arms: 1
Dietary Supplement: Lactobacillus acidophilus NCFM — 1e10 CFU/day
  Arms: Active 1
Dietary Supplement: Combination of Lactobacillus acidophilus and Bifidobacterium lactis — 1x10e10 CFU/day
  Arms: Active 2

SUMMARY:
The aim of the present prospective study is to investigate whether the consumption of certain probiotic strains over a six-month winter/spring season would be able to affect the incidence and duration of upper respiratory tract infections, in otherwise healthy children as well as determining whether a combination of two strains would perform differently from a single strain version.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-5 years of normal nutritional status and health

Exclusion Criteria:

* Contraindications to dairy products (lactose intolerance or cow's milk allergy)
* Indicators of inflammatory disease, intestinal disease, Crohn's disease, colitis, celiac disease
* Chronic cough from recurring respiratory distress-related diseases
* Hirschsprung's disease
* Cystic fibrosis
* Other metabolic, neurological, or anatomic alteration that predisposes participation
* Intake of probiotics within the last 3 weeks

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 326 (Actual)
Dates: Start 2005-11; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To examine if the consumption of two different probiotic strains added to milk at the point of consumption could reduce the "flu-like" symptoms and other symptoms of illness of preschool-age children in day care centers. | Daily for six months

SECONDARY OUTCOMES:
To determine if children who consume a beverage fortified with a probiotic miss fewer days of preschool as measured by illness. | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Zhang, Study Director — Sprim Advanced Life Sciences; Cheryl Riefer, Study Chair — Sprim Advanced Life Sciences
Locations (1):
- Day care center, Jinhua, Zhejiang, China

REFERENCES:
- [Derived] Leyer GJ, Li S, Mubasher ME, Reifer C, Ouwehand AC. Probiotic effects on cold and influenza-like symptom incidence and duration in children. Pediatrics. 2009 Aug;124(2):e172-9. doi: 10.1542/peds.2008-2666. Epub 2009 Jul 27. PMID 19651563